CLINICAL TRIAL: NCT01494363
Title: Multicenter Phase II Study of Fluorouracil, Leucovorin, Oxaliplatin, and Irinotecan (FOLFOXIRI) in Patients With Locally Advanced or Metastatic Biliary Tract Cancer
Brief Title: Phase II Study of FOLFOXIRI in Patients With Locally Advanced or Metastatic Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Nam Su Lee, Professor, Soon Chun Hyang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCH01
Record Dates: First submitted 2011-12-13; First posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Fluorouracil — 5-fluorouracil 2400 mg/m2 (diluted in 1000 ml of 5% dextrose solution) administered as a continuous intravenous infusion over 48 hours every 2 weeks
Drug: Leucovorin — Leucovorin 400 mg/m2 (diluted in 250 ml of 5% dextrose solution) as a 2-hour intravenous infusion every 2 weeks
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2 (diluted in 250 ml of 5% dextrose solution) given as a 2-hour intravenous infusion every 2 weeks
Drug: Irinotecan — Irinotecan 150 mg/m2 (diluted in 250 ml of 0.9% normal saline solution) given as a 90-minute intravenous infusion every 2 weeks

SUMMARY:
1. Goals

   The primary goal of this phase II trial is to:

   evaluate the response rate of combination chemotherapy with Fluorouracil, Leucovorin, Oxaliplatin, and Irinotecan in patients with locally advanced or metastatic Biliary tract cancer as first-line chemotherapy

   Secondary goals are to:

   evaluate the treatment-related toxicities of this combination, investigate progression-free survival(PFS) and overall survival(OS) in this population
2. Design The proposed clinical trial is an open label, non-comparative, multicenter phase II trial according to the two stage testing design by Simon two-stage testing procedure

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed as adenocarcinoma of gallbladder or biliary tract histologically or cytologically
2. Unresectable locally advanced, metastatic, or recurrent biliary tract cancer
3. Patients must be ≥ 18 , ≤ 75 years old of age
4. ECOG performance status ≤ 2
5. At least one lesion that can be measured by imaging (CT/MRI) according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
6. Estimated life expectancy of more than 3 months
7. Adequate bone marrow function (absolute neutrophil count [ANC] ≥ 1,500/µL, hemoglobin ≥ 9.0 g/dL [correction by transfusion is acceptable], and platelets ≥ 100,000/µL)
8. Adequate kidney function (serum creatinine < 1.5 x upper limit of normal [ULN])
9. Adequate liver function (serum total bilirubin < 3.0xULN; serum transaminases levels < 5.0xUNL)
10. Provision of fully informed consent prior to any study specific procedures

Exclusion Criteria:

1. Other tumor type than adenocarcinoma
2. Any previous history of chemotherapy for biliary tract cancer (prior neoadjuvant/adjuvant chemotherapy is allowed, if recurrence occurred more than 6 months after completion of previous chemotherapy)
3. Patients with second primary cancer (except, adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥5 years)
4. Patients who received radiotherapy on target lesion within 6 months prior to study treatment
5. Patients with defect of central nervous system (CNS) or any psychiatric disorders and CNS metastases
6. Patients who received major surgery within 4 weeks of starting study treatment or was not recovered from any effects of major surgery
7. Pregnant or breastfeeding women and women of childbearing potential not employing adequate contraception
8. Other serious illness or medical conditions A. Clinically significant cardiac disease (uncontrolled congestive heart disease despite treatment [NYHA class III or IV], symptomatic coronary artery disease, unstable angina or myocardial infarction, conduction abnormality like grade 2 AV block, serious arrhythmia needed for medication, uncontrolled hypertension) within 6 months prior to study entry B. Liver cirrhosis (≥ Child-Pugh class B) C. History of significant neurologic or psychiatric disorders including dementia or seizures D. Active uncontrolled infection E. Other serious underlying medical conditions which could impair the ability of the patient to participate in the study
9. Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 2 years
  Assessment of response will be assessed according to RECIST v1.1 criteria after completion of every two cycles. Evaluation will be conducted by physical examination, X-ray, or CT scan

SECONDARY OUTCOMES:
Treatment-related toxicities | 2 years
  Assessment of toxicity will be assessed according to NCI CTCAE version 4.0.
Progression free survival | 2 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Hyun Jung Kim, Bucheon-si
  - Han Jo Kim, Cheonan
  - Nam Su Lee, Seoul